CLINICAL TRIAL: NCT03001856
Title: Interrupted Oblique Intradermal Suture Versus Conventional Interrupted Intradermal Suture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Apinut Wongkietkachorn, Doctor, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MaeFahLuangUH
Record Dates: First submitted 2016-12-19; First posted 2016-12-23 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oblique Intradermal Suture (Experimental): OIS is very similar to conventional interrupted intradermal suture (IS), except that the suture in OIS is canted or angled relative to the vertical plane (Figure 1). To perform OIS, the needle is passed from deep to superficial dermis and canted 30°-60° from the normal vertical plane. The needle is then inserted into the opposite wound edge from superficial to deep dermis in a mirror-image fashion. The thread is tied with a square knot to finish the suture.
  Interventions: Procedure: Oblique Intradermal Suture
- Intradermal Suture (Experimental): Conventional interrupted intradermal suture
  Interventions: Procedure: Intradermal Suture

INTERVENTIONS:
Procedure: Oblique Intradermal Suture
  Arms: Oblique Intradermal Suture
Procedure: Intradermal Suture
  Arms: Intradermal Suture

SUMMARY:
This study was conducted to demonstrate the equivalence of wound outcomes between the interrupted oblique intradermal suture (OIS) and conventional interrupted intradermal suture (IS) methods

DETAILED DESCRIPTION:
Bi-layered skin closure is one of the most common methods for closing cutaneous defects. The deep layer is closed with a conventional interrupted intradermal suture using absorbable materials, while the superficial layer is approximated with simple interrupted or simple continuous suture using non-absorbable materials. The cosmetic result of bi-layered closure is better than simple interrupted suture alone, because the interrupted intradermal suture component plays a major role in reducing wound tension, which has the effect of minimizing suture marks. Although the advantages of bi-layered closure are recognized, bi-layered closure is often not used in favor of simple interrupted suture due to the fact that interrupted intradermal suture is time consuming and more suture material is required. Thus, if an intradermal suturing technique can be identified that takes less time and requires less material while yielding a similar cosmetic result, patients would have more opportunity to receive bi-layered closure and obtain a better wound outcome.

Several novel intradermal suturing techniques could be alternative to the conventional interrupted intradermal suture technique, including buried butterfly suture, double butterfly suture, subcutaneous inverted cross mattress suture, and interrupted oblique intradermal suture. Among these novel techniques, interrupted oblique intradermal suture (OIS) is recognized for its relative simplicity. OIS is easy to perform, even for beginners. The simplicity and effectiveness of OIS increase its potential of becoming one of the standard suturing techniques in medical practice.

OIS is very similar to conventional interrupted intradermal suture (IS), except that the suture in OIS is canted or angled relative to the vertical plane. To perform OIS, the needle is passed from deep to superficial dermis and canted 30°-60° from the normal vertical plane. The needle is then inserted into the opposite wound edge from superficial to deep dermis in a mirror-image fashion. The thread is tied with a square knot to finish the suture. The key characteristic that distinguishes OIS from IS is that OIS involves suturing on an angle to the vertical plane and IS involves suturing on the vertical plane.

In theory, OIS is a hybrid method that combines IS and buried horizontal butterfly suture. OIS combines the ability of IS to reduce tension at the wound edge and the ability of horizontal butterfly suture to provide good wound edge apposition and eversion. Because OIS is canted, it can provide tension in both the vertical and horizontal planes. Moreover, 1 stitch of OIS should yield wound closure approximately equal to that of 2 stitches of IS due to the same horizontal distance between 1 OIS stitch and 2 VIS stitches. Accordingly, it can be inferred that OIS should result in a 50% reduction in both suturing time and suturing material used.

However, OIS has the same obstacle as many other novel suturing techniques that there is very little literature to support OIS clinically which makes usage and generalization of TIS remain limited. It was hypothesized that OIS is equivalence to IS in wound outcome while consumes less time and less suture material. This study aims to demonstrate the equivalence of wound outcomes between the interrupted oblique intradermal suture (OIS) and conventional interrupted intradermal suture (IS) methods.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* needs elective surgery with linear incision wound
* wound length must be 3-12 cm.

Exclusion Criteria:

* irregular wound shape
* asymmetrical wound depth
* different skin color in wound area
* contaminated wound
* mental impairment
* pregnancy
* patients with soft tissue disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Modified Hollander Cosmesis Scale (MHCS) at 1st week | 1 week
  Wound evaluation at 1st week
Patient and Observer Scar Assessment Scale (POSAS) at 1st week | 1 week
  Wound evaluation at 1st week
Modified Hollander Cosmesis Scale (MHCS) at 2nd month | 2nd month
  Wound evaluation at 2nd month
Patient and Observer Scar Assessment Scale (POSAS) at 2nd month | 2nd month
  Wound evaluation at 2nd month

SECONDARY OUTCOMES:
Rate of wound dehiscence | 1 week
Rate of wound infection | 1 week
Suture time | day 1
Number of stitches | day 1
Suture material length | day 1

REFERENCES:
- [Derived] Wongkietkachorn A, Wongkietkachorn N, Rhunsiri P. Oblique intradermal suture as a faster choice for intradermal closure: a randomized equivalence trial. J Plast Surg Hand Surg. 2019 Feb;53(1):45-50. doi: 10.1080/2000656X.2018.1533476. Epub 2018 Oct 31. PMID 30380956